CLINICAL TRIAL: NCT05138224
Title: Is There a Higher Prevalence of Autistic Spectrum Disorder (ASD) in Children With Haemophilia (Aged 5-16) Than the General Population?
Brief Title: Prevalence of Autistic Spectrum Disorder (ASD) in Children With Haemophilia
Status: Completed | Type: Observational
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 10MH17
Record Dates: First submitted 2020-11-25; First posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Haemophilia; Autism Spectrum Disorder; Social Communication Disorder; Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Hemophilia A; Autism Spectrum Disorder; Social Communication Disorder; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Parents of children with haemophilia will be invited to complete 3 questionnaires to look for traits present in ASD. With consent teacher will complete a further 2 questionnaires. If all 3 questionnaires are above threshold, then with consent of the family the child will be referred for further investigation.

There are already pre-existing children with ASD who will be exempt from the study, but included in the data analysis of prevalence.

The results of the 3 questionnaires will be used to identify a profile of social communication in children with haemophilia.

DETAILED DESCRIPTION:
Background Haemophilia A and B are inherited disorders characterised by spontaneous bleeding. The current treatment is replacement of the deficient factor VIII (FVIII) or factor IX (FIX). Haemophilia occurs in 1:50000 male births and approximately 85% have haemophilia A and approx 15% haemophilia B. Children with haemophilia can be described as having severe, moderate or mild disease dependent on their circulating levels of FVIII or FIX. Children with severe haemophilia are classified as having <1%, moderate 1-5% and mild >5-40%. One third of all children diagnosed with haemophilia have no family history of the bleeding disorder. 80% of bleeding episodes occur in the joints. A bleed into the cranial cavity although rare is called an intracranial haemorrhage (ICH) and outcome can range from neurological impairment (behavioural difficulties) to death (1-2). Bladen et al. 2009 identified behavioural difficulties in a cohort of children at Great Ormond St Hospital for Children NHS Trust with haemophilia following intracranial haemorrhage (3).

Haemophilia and communication difficulties A recent study has highlighted that boys with haemophilia risk attention deficit / hyperactivity disorder (ADHD) spectrum difficulties especially hyperactivity impulsivity (HI) and special education participation (4). No papers could be found detailing a relationship or prevalence of autistic spectrum disorder and haemophilia.

Since the Bladen et al. 2009 publication there has been an increased awareness and diagnosis of boys with autistic spectrum disorder (ASD) at Great Ormond St Hospital for Children NHS Trust haemophilia centre. These problems have required the children to gain statements of special education need in order that they can maximise their educational potential. Children with ASD can also present with motor co-ordination difficulties that increase their risk of falls. This tendency to lack control of their movement may increase bleeding frequency in boys with haemophilia placing them at further risk. It is essential that these boys are screened and identified early so that the necessary additional these children require is attained.

Current literature states that ASD affects approximately 1% of the general population (5-6). Autism-spectrum disorders are diagnosed by the presence of social and communication difficulties, alongside unusually strong, narrow interests and/or repetitive and stereotyped behaviour (7). Language delay and difficulties in cognitive ability are common in children and may extend into below-average range intellectual disabilities. For clinical purposes diagnosis is set at the level where autistic traits are significantly interfering in daily life functioning; currently, there is no biological marker and the diagnosis is established on a basis of a comprehensive assessment of children's behavioural characteristics.

Aim of the study The aim of this study is to use questionnaires to be completed by parents and teachers to screen and assess for difficulties in social interactions, executive functioning, communication and behaviour in boys with haemophilia aged 5-16 .

This research will establish if there is a higher prevalence of symptoms of ASD and executive function difficulties in boys with haemophilia than the general population. This knowledge will assist education management strategies to help those affected boys maximise their educational potential through appropriate schooling support. Highlighting ASD symptoms may aid early diagnosis and facilitate earlier management strategies e.g. a statement of special of educational need if required. The proposed study intends to identify if the increased number of children we have with ASD is an artefact or if indeed there is a higher prevalence of ASD in children with haemophilia. If these findings are substantiated then in the future all children with haemophilia will be screened for ASD as appropriate. Children with above threshold scores on all 3 questionnaire scores would then be referred locally for further psychological assessment and possible diagnosis . All children referred locally for further psychological assessment will be followed up to ascertain if a diagnosis is made as per routine clinical practice. An earlier diagnosis would hopefully ensure that the child and family receive earlier support and maximise the child's potential. It is anticipated that the completion of this study will help improve the overall care and management of boys with haemophilia and autistic spectrum disorder.

Methodology Subjects aged 5-16 years with haemophilia will be identified from Great Ormond St hospital for children NHS Trust haemophilia database. Subjects less than 5 years of age, over 16 years of age, with other bleeding disorders or those already with a diagnosis of ASD will be excluded. The study population is parents of boys with a diagnosis of haemophilia aged 5-16 years of age. It is hoped there will be 100 eligible subjects to take part as the total cohort is 149. Parents of children aged 5-16 years of age will be contacted by letter two weeks before their scheduled haemophilia review (see attached) to invite them to participate in the questionnaire research and they will also be provided with an information leaflet with the invite On attendance at the haemophilia centre if the family agree to participate, consent will be obtained (see attached Parent consent form). This will include consent to contact the child's head teacher, class teacher and the G.P. It is acknowledged that parents may experience increased anxiety whether their child has problems or not and as such it is essential the GP is aware of the family's participation in this study.

For those parents who are unable to read or speak English an interpreter will be provided. Arrangement of an interpreter would be pre-booked for their review appointment as normal. Completion of the form shall be assisted by another member of the team.

Once consent has been obtained, the child's head teacher and class teacher will be contacted with a letter along with a teachers information sheet (see attached) and a copy of the signed consent form. This will inform them of the study and invite them to participate. The class teacher should have known the child for more than 3 months As well as the questionnaires additional information will be gathered from the medical notes and parents, such as birth history, current medication, educational status e.t.c.(for all the items please see attached Additional information sheet) The following questionnaires have been shown to be reliable and valid for screening for children with ASD, The Social Communication Questionnaire, The Childrens Communication Checklist (CCC-2) and the Behaviour Rating Inventory of Executive Function (BRIEF). All questionnaires have normative data for comparison and as such a control group is not required. These 3 will be completed by the parent on the day of the assessment, whilst their child is receiving their routine musculoskeletal assessment. The BRIEF and CCC questionnaires will be sent with the teachers invitation for them to complete. A follow up telephone call will be made to the teacher to discuss any questions they may have .

The Social Communication Questionnaire (SCQ) (8) The SCQ is a brief instrument that can be used to evaluate children over 4 years of age as long as his or her mental age exceeds 2 years of age. The questionnaire takes approximately 10-15 minutes to complete. The questionnaire focuses on behaviours that are rare in non-affected individuals and can be used as a screener for autistic spectrum disorder.

The Social Communication Questionnaire is a 40 item yes/no response parent-report questionnaire that asks about characteristic autistic behaviour. There are 2 forms; the autoscore looking at behaviour in the last 3 months and the lifetime score. The total score is a combination of the autoscore and lifetime score and is interpreted in relation to cut-off scores that indicate the likelihood of an individual having ASD.

The items are scored as either 0 or 1. A score of 1 is an endorsement for each symptom of autism. The range of scores is from 0-39 as the first item the language score is not included in the total score. Nineteen items rate current behaviour and 20 rate behaviour when the child was 4-5 years old. The recommended cut-off score for autistic-spectrum disorder or pervasive developmental disorder is >15. The SCQ has been found to have a high discriminant ability in differentiating ASD symptomatology from other associated behavioural and developmental difficulties. (9).

The Behaviour Rating Inventory of Executive Functioning (BRIEF) (10) Executive functioning is a collection of functions that are responsible for guiding, directing and managing cognitive, emotional and behavioural functions particularly during active, novel problem solving. The term executive function is an umbrella term to describe a collection of inter-related functions that are responsible for purposeful, goal directed problem-solving behaviour.

The BRIEF questionnaire is for parents and teachers of school-aged children that enables professionals to assess executive functioning at home and in the school environments. Answering if any of the statements have applied to the child in the past 6 months. It is designed for children aged 5-18 years of age, and recommended for use with children with a wide range of developmental and neurological conditions, such as ADHD and ASD, who have been identified to be at an increased risk of possible executive function difficulties, including those with learning disabilities, attentional disorders and brain injuries. The questionnaire will take 10- 15 minutes to complete.

The BRIEF contains 86 items within eight theoretically and empirically derived clinical scales that measure and monitor different aspects of executive functioning: inhibit, shift, emotional control, initiate, working memory, plan/organise, organisation of materials.

Inhibit - Assesses inhibitory control i.e. the ability to inhibit, resist or not act on ones impulses.

Shift- Assesses the ability to move freely from one situation or activity or aspect of a problem to another as circumstances demand (problem solving).

Emotional control - Assesses the ability to modulate emotional control i.e. emotional lability or emotional explosiveness.

Initiate - Assesses items relating to beginning a task or activity as well as independently generating ideas, responses or problem solving strategies.

Working memory - Assesses the capacity to hold on to information in mind for the purpose of completing a task. Working memory is essential to carry out multistep activities, complete mental arithmetic or follow complex instructions.

Plan / organise - Assesses the child's ability to manage current and future-orientated tasks. The plan element takes in to consideration an ability to anticipate future events, set goals and set appropriate steps to complete the task. The organise component involves assessing written and oral information to bring order to information and to appreciate the main ideas or concepts.

Organisation of materials - Assesses a child's orderliness of work, play and storage space. This may also take into consideration how order is brought about.

The BRIEF has been shown to have good reliability and validity (10-11). The Childrens Communication Checklist (CCC-2) (12-13) This questionnaire is a 70 item questionnaire which has standard scores and percentiles and can be completed by the parent or teacher The questionnaire asks about language and communication. Scoring an item is broken down into 0 ('does not apply'), 1 ('applies somewhat'), 2 ('definitely applies') or missing value ('unable to judge'). This questionnaire will take approximately 10-15 minutes to complete.

The CCC-2 is divided into 9 subscales: two sub-scales assess aspects of language structure (syntax and speech); two assess aspects of autistic behaviour (social relationships and interests); and five assess aspects of pragmatic communication (inappropriate initiation, coherence, stereotyped conversation, use of context, and rapport), which has been found to be impaired in children with ASD. The raw scores of the subscales are converted to aged scaled scores with a mean of 10 and a std of 3. These aged scaled scores and the GCC are converted to percentiles.

The CCC-2 (12) has a pragmatic composite sub-scale that has been shown to distinguish between those individuals with and without autistic spectrum disorder (14). The CCC-2 has been used in the literature to identify children with communication impairments from non-impaired peers (15). (See attached for copies of the questionnaires proposed) The supervision and scoring of these questionnaires shall be undertaken by Marianna Murin, Clinical Psychologist who works in the social communication team at Great Ormond Street Hospital for Children NHS Trust. The supervision will consist of an initial training session, followed by observed practical sessions. The administration of the questionnaires will be carried out by the primary investigator and Nicola Hubert Physiotherapy colleague.

A score on a screening instrument is indicative of a probable Autism Spectrum Disorder, however it is not sufficient for a formal diagnosis. For diagnostic assessment a full parental interview regarding current and past development and behaviour, and structured observation of the child, preferably including a peer-group setting, is essential. Those children with questionnaire results that suggest further assessment is required will be discussed with Marianna Murin. The family shall be informed by telephone of the concerns raised from the assessment, either by Marianna Murin, the primary investigator or Nicola Hubert physiotherapy colleague. The report will be written and sent to the family. In consultation and consent with the family a referral to a local psychologist via the GP or local paediatrician will be made to facilitate further assessments and establish a diagnosis along with appropriate intervention and support. In the unlikely event of a lost referral / lost letter the primary investigator will follow up all children referred to local services to ensure the referral is received and the outcome of their assessments is known. This would follow current clinical practice. Those children with no indication for ongoing assessment will not receive a report, but a letter that states there is no indication for further investigation.

Results The time scale from invitation to receipt of a letter detailing the outcome of the assessment shall take approximately 6 weeks.

Analyses of the results have been discussed with Angie Wade in the Institute of Child Health.

Previous research within the haemophilia unit has demonstrated a high rate of return with this population group and as such a 5-10% drop out rate is typical of previous studies.

The power calculation provided has considered that some individuals may decline to participate. Based on a sample of 140 out of 149 subjects, we expect at-least 10% to test positive. We would estimate this to + or - 5%. At most we anticipate 33% testing positive and in this case the precision would be + or - 8%. Therefore the sample provides sufficient precision.

The overall results of the study shall be published in a peer review journal. A summary of the overall findings shall be published in the Great Ormond Street Hospital for Children NHS Trust Haemophilia Centre newsletter that is distributed to all families with a child with haemophilia.

Duration of study It is anticipated that data collection will take 1 year and will start in January 2013 and be completed January 2014. Data analysis should be completed by July 2014.

ELIGIBILITY:
Inclusion Criteria:

-All boys with mild, moderate or severe haemophilia will be offered to participate in the questionnaire completion

Exclusion Criteria:

-boys with a pre-existing diagnosis of ASD will be excluded from questionnaire completion but will be included in the prevalence analysis

Ages: 5 Years to 16 Years | Sex: Male
Age Groups: Child
Gender Based: Yes — All boys with haemophilia at Great Ormond St Hospital haemophilia centre
Study Population: All boys with all severities of haemophilia aged 5-16 years
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2014-09; Primary Completion 2018-08 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of autism spectrum disorder in boys with haemophilia at Great Ormond St Hospital | Within 2 weeks of when the participant consented- measured once
  The number of children with a diagnosis of ASD at GOSH

SECONDARY OUTCOMES:
Social Communication Questionnaire | Within 2 weeks of when the participant consented-measured once
  Questionnaire Scores > or equal to 15 will be considered positive
Childrens communication Checklist | Within 2 weeks of when the participant consented-measured once
  Questionnaire Scores < or equal to 132 will be considered positive
BRIEF | Within 2 weeks of when the participant consented-measured once
  Questionnaire Scores on the global executive composite score of > or equal to 65 will be considered positive
Number of children being given a diagnosis of ASD or other following referral for ongoing assessment following positive scores on questionnaires | From when study started October 2014 to study end July 2017
  Children gaining above threshold on the SCQ, CCC and BRIEF and with consent of the family will be referred locally, assessed and the number of children gaining an additional diagnosis will be recorded

REFERENCES:
- [Background] Kulkarni R, Lusher JM. Intracranial and extracranial hemorrhages in newborns with hemophilia: a review of the literature. J Pediatr Hematol Oncol. 1999 Jul-Aug;21(4):289-95. doi: 10.1097/00043426-199907000-00009. PMID 10445891
- [Background] Ljung RC. Intracranial haemorrhage in haemophilia A and B. Br J Haematol. 2008 Feb;140(4):378-84. doi: 10.1111/j.1365-2141.2007.06949.x. Epub 2007 Dec 13. PMID 18081890
- [Background] Bladen M, Khair K, Liesner R, Main E. Long-term consequences of intracranial haemorrhage in children with haemophilia. Haemophilia. 2009 Jan;15(1):184-92. doi: 10.1111/j.1365-2516.2008.01815.x. Epub 2008 Aug 13. PMID 18702617
- [Background] Spencer ML, Wodrich DL, Schultz W, Wagner L, Recht M. Inattention, hyperactivity-impulsivity, academic skills and psychopathology in boys with and without haemophilia. Haemophilia. 2009 May;15(3):701-6. doi: 10.1111/j.1365-2516.2009.01993.x. Epub 2009 Feb 27. PMID 19298375
- [Background] Baird G, Simonoff E, Pickles A, Chandler S, Loucas T, Meldrum D, Charman T. Prevalence of disorders of the autism spectrum in a population cohort of children in South Thames: the Special Needs and Autism Project (SNAP). Lancet. 2006 Jul 15;368(9531):210-5. doi: 10.1016/S0140-6736(06)69041-7. PMID 16844490
- [Background] Baron-Cohen S, Scott FJ, Allison C, Williams J, Bolton P, Matthews FE, Brayne C. Prevalence of autism-spectrum conditions: UK school-based population study. Br J Psychiatry. 2009 Jun;194(6):500-9. doi: 10.1192/bjp.bp.108.059345. PMID 19478287
- [Background] Chandler S, Charman T, Baird G, Simonoff E, Loucas T, Meldrum D, Scott M, Pickles A. Validation of the social communication questionnaire in a population cohort of children with autism spectrum disorders. J Am Acad Child Adolesc Psychiatry. 2007 Oct;46(10):1324-1332. doi: 10.1097/chi.0b013e31812f7d8d. PMID 17885574
- [Background] Offord DR, Boyle MH, Racine Y, Szatmari P, Fleming JE, Sanford M, Lipman EL. Integrating assessment data from multiple informants. J Am Acad Child Adolesc Psychiatry. 1996 Aug;35(8):1078-85. doi: 10.1097/00004583-199608000-00019. PMID 8755805
- [Background] Bishop DV. Development of the Children's Communication Checklist (CCC): a method for assessing qualitative aspects of communicative impairment in children. J Child Psychol Psychiatry. 1998 Sep;39(6):879-91. PMID 9758196
- [Background] Bishop DV, Baird G. Parent and teacher report of pragmatic aspects of communication: use of the children's communication checklist in a clinical setting. Dev Med Child Neurol. 2001 Dec;43(12):809-18. doi: 10.1017/s0012162201001475. PMID 11769267
- [Background] Norbury CF, Nash M, Baird G, Bishop D. Using a parental checklist to identify diagnostic groups in children with communication impairment: a validation of the Children's Communication Checklist--2. Int J Lang Commun Disord. 2004 Jul-Sep;39(3):345-64. doi: 10.1080/13682820410001654883. PMID 15204445
- [Background] World Health Organization. The ICD-10 Classification of Mental and Behavioural Disorders: Diagnostic Criteria for Research. WHO, 1993.
- [Background] Rutter, M., Bailey, A. & Lord,C. (2003) Social Communication Questionnaire (SCQ).Western Psychological Services.
- [Background] Gioia, G.A., Isquith, P.K., Guy, S.C., Kenworthy, L. (2000) Behaviour rating inventory of executive functioning Florida: Psychological Assessment Resources Inc.
- [Background] Bishop DVM. (2003) Children's Communication Checklist Version 2 (CCC2). Psychological Corporation.